CLINICAL TRIAL: NCT07014657
Title: Effect of Digital Combined Decongestive Therapy in Patients With Breast Cancer-related Lymphedema: a Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Selva Otsay, Principal Investigator, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lenfödemüst2025
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer-Related Lymphedema
Keywords: Breast cancer-related lymphedema; Combined decongestive therapy; Digital therapy
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Combined Decongestive Therapy Group (Experimental): Participants received digital combined decongestive therapy including self-bandaging, self-manual lymphatic drainage, decongestive and breathing exercises, supervised remotely through telecommunication technologies for 4 weeks, followed by maintenance therapy with compression stockings.
  Interventions: Behavioral: Digital Combined Decongestive Therapy

INTERVENTIONS:
Behavioral: Digital Combined Decongestive Therapy — Participants received digital combined decongestive therapy, which included an initial face-to-face session where skin care and risk reduction training were provided. Self-bandaging and self-manual lymphatic drainage techniques were demonstrated and practiced under supervision. Additionally, decongestive and breathing exercises were taught to both patients and caregivers. Following this, the intensive treatment phase was conducted remotely using electronic communication technologies over a period of 4 weeks to monitor and guide the therapy. After the intensive phase, participants continued with maintenance therapy, which involved the use of compression stockings. The therapy aimed to reduce limb volume and improve symptoms related to breast cancer-related lymphedema.

SUMMARY:
This study investigated the short- and long-term effects of digital combined decongestive therapy in breast cancer-related lymphedema. Limb volume and quality of life (Lymph-ICF) were assessed at baseline, post-treatment, and 12-week follow-up.

DETAILED DESCRIPTION:
This study evaluated the feasibility and effectiveness of a digital combined decongestive therapy (CDT) program in patients with breast cancer-related lymphedema. After an initial face-to-face training session on self-bandaging, self-manual lymphatic drainage, breathing exercises, and skin care, patients followed a 4-week digital CDT program with remote guidance. Compression garments were used during the maintenance phase. Limb volume was measured using circumference method. Quality of life was assessed with the Lymph-ICF questionnaire. Assessments were repeated post-treatment and at 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer-related lymphedema (BCRL) within the last 6 to 60 months.
* Voluntarily agreed to participate in the study.

Exclusion Criteria:

* Presence of active infection.
* History of bilateral breast surgery.
* Severe breast cancer-related lymphedema.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Limb Volume | At baseline, at week 4 (end of treatment), and at week 12 (follow-up)
  Limb volume was assessed by measuring the circumference of the affected arm at 4-cm intervals from the ulnar styloid to the axillary region using a standard tape measure. These measurements were used to calculate the total limb volume to evaluate changes after the intervention and at follow-up.

SECONDARY OUTCOMES:
Change in Quality of Life | At baseline, at week 4 (end of treatment), and at week 12 (follow-up)
  Quality of life was assessed using the Turkish validated and reliable lymphedema-specific questionnaire, Lymph-ICF. The questionnaire consists of 29 items including 7 questions about arm symptoms and 22 questions related to functional impairments in daily activities. It covers five subscales: physical function, mental status, household activities, mobility activities, and social life. Patients rated their complaints on a 0 to 100 mm visual analog scale (VAS), where 0 indicates no complaints and 100 indicates the worst complaints. Higher scores represent worse quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borman P, Yaman A, Yasrebi S, Pinar Inanli A, Arikan Donmez A. Combined Complete Decongestive Therapy Reduces Volume and Improves Quality of Life and Functional Status in Patients With Breast Cancer-Related Lymphedema. Clin Breast Cancer. 2022 Apr;22(3):e270-e277. doi: 10.1016/j.clbc.2021.08.005. Epub 2021 Aug 19. PMID 34535391